CLINICAL TRIAL: NCT04373720
Title: Pilot Study to Assess Mean Lesion Stiffness of Radiation Necrosis and Recurrent Glioma Using Magnetic Resonance Elastography (MRE) in Patients With Previously Treated Gliomas
Brief Title: MRE Scan for the Assessment of Differences in Tissue Stiffness Between Radiation Necrosis and Recurrent Glioma in Patients With Previously Treated Gliomas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-1070; NCI-2020-02247 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1070 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (MRE, standard of care MRI) (Experimental): Patients undergo MRE over 10 minutes and then undergo standard of care MRI of the brain with and without contrast at baseline. Within 4 weeks after the initial MRI and MRE scans, patients may undergo standard of care biopsy to check the status of the disease. Within 48 hours after biopsy, patients undergo standard of care MRI to check the status of the disease. Patients who do not undergo biopsy undergo standard of care MRI 4-8 weeks after MRE scan to check the status of the disease.
  Interventions: Procedure: Magnetic Resonance Elastography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Magnetic Resonance Elastography — Undergo MRE
  Other Names: MRE
Procedure: Magnetic Resonance Imaging — Undergo standard of care MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This trial uses magnetic resonance elastography (MRE) to estimate tissue stiffness (hardness or softness of the tissue) in tissue that is affected by radiation treatment (radiation necrosis) and tumor tissue that has come back (recurrent) after treatment in patients with gliomas. Diagnostic procedures, such as MRE, may estimate the differences in tissue stiffness between radiation necrosis and recurrent glioma post treatment and ultimately lead to a more accurate diagnosis and/or surgery, and/or a better assessment of the disease's response to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the mean lesion stiffness in patients with radiation necrosis using magnetic resonance elastography (MRE).

II. To estimate the mean lesion stiffness in patients with glioma recurrence using magnetic resonance elastography (MRE).

SECONDARY OBJECTIVE:

I. To investigate the mean lesion stiffness between radiation necrosis and glioma recurrence.

OUTLINE:

Patients undergo MRE over 10 minutes and then undergo standard of care magnetic resonance imaging (MRI) of the brain with and without contrast at baseline. Within 4 weeks after the initial MRI and MRE scans, patients may undergo standard of care biopsy to check the status of the disease. Within 48 hours after biopsy, patients undergo standard of care MRI to check the status of the disease. Patients who do not undergo biopsy undergo standard of care MRI 4-8 weeks after MRE scan to check the status of the disease.

ELIGIBILITY:
Inclusion Criteria

* >/=18 years old.
* History of a pathology proven intracranial glioma (including IDH mutant, IDH wildtype or 1p19q co-deleted tumors) treated with chemotherapy and radiation.
* The lesion of concern (T2 Flair Hyperintense or contrast enhancing lesion) is > 2 cm
* Patient is able to understand and give consent to participation in the study.

Exclusion Criteria

* Patients less than 18 years of age.
* Pregnant.
* Known allergy to gadolinium-based contrast agents.
* Renal failure as evidenced by a glomerular filtration rate (GFR) of less than 30 mL/min/1.73m2.
* Pacemakers, electronic stimulation, metallic foreign bodies and devices and/or other conditions that are not MR safe, which include but are not limited to:

  * electronically, magnetically, and mechanically activated implants
  * ferromagnetic or electronically operated active devices like automatic cardioverter defibrillators and cardiac pacemakers
  * metallic splinters in the eye
  * ferromagnetic hemostatic clips in the central nervous system (CNS) or body
  * cochlear implants
  * other pacemakers, e.g., for the carotid sinus
  * insulin pumps and nerve stimulators
  * non-MR safe lead wires
  * prosthetic heart valves (if dehiscence is suspected)
  * non-ferromagnetic stapedial implants
  * claustrophobia that does not readily respond to oral medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Mean lesion stiffness | At baseline
  For each patient, a lesion region of interest (ROI) will be created along with its normal appearing contralateral white matter. The stiffness of the tumor ROI and the contralateral white matter ROI will be measured, and the ratios of the stiffness between the two will be calculated. Interval estimates will be computed for mean stiffness ratio in patients with radiation necrosis or glioma recurrence, separately using a 2-sided 95% confidence interval. Outcome variable of stiffness will be assessed between tumor and contralateral white matter with paired t-tests or Wilcoxon signed-rank tests. The Wilcoxon rank-sum test or t-tests will be used to assess the associations between the outcome variable of stiffness ratio and tumor status (recurrence/necrosis).

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Chen, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org